CLINICAL TRIAL: NCT04325152
Title: Clip-assisted Fixation to Prevent Migration of Fully Covered Self-expandable Metal Stent in Patients Undergoing ERCP: a Randomized Controlled Trial
Brief Title: Clip-assisted Fixation to Prevent Migration of Fully Covered Self-expandable Metal Stent in Patients Undergoing ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Huaihe Hospital of Henan University (Other); Xiamen Humanity Hospital (Other); The Third Affiliated Hospital of Second Military Medical University (Unknown)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY20200113-2
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Pancreaticobiilary Diseases; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; Fully Covered Self-expandable Metal Stent
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCSEMS+Clip (Experimental): After successful cannulation, a 10mm FCSEMS with the length of 6cm or 8cm were inserted into CBD. One to two centimeters of distal end of FCSEMS was left outside of the papilla and the stent was released. Then a metal clip was used to fix the distal end of FCSEMS with the duodenal mucosa adjacent to papilla.
  Interventions: Device: FCSEMS plus Clip
- FCSEMS (Sham Comparator): FCSEMS was released as the same as mentioned above. No fixating method was used.
  Interventions: Device: FCSEMS

INTERVENTIONS:
Device: FCSEMS plus Clip — After successful cannulation, a 10mm FCSEMS with the length of 6cm or 8cm were inserted into CBD. Then a metal clip was used to fix the distal end of FCSEMS with the duodenal mucosa adjacent to papilla.
  Arms: FCSEMS+Clip
Device: FCSEMS — FCSEMS was released as the same as mentioned above. No fixating method was used.
  Arms: FCSEMS

SUMMARY:
Fully covered self-expandable metal stent (FCSEMS) has been widely used in ERCP patients with malignant or benign biliary stricture, difficult CBDS, post-EST bleeding, bile leak or perforation. Compared with uncovered SEMS, FCSEMS can be removed several months later and has the advantage of longer patency. Proximal or distal migration is one of major disadvantages of FCSEMS. The migration rate ranged from 7.0%-33% in previous reports.

We hypothesized that the fixation of the distal end of FCSEMS by a metal clip could decrease the migration rate and migration-related cholangitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Patients with ERCP indications who were suitable for FCSEMS placement, such as benign or malignant biliary stricture, difficult CBDS, biliary or papillary bleeding, bile leak or perforation etc.

Exclusion Criteria:

1. Expected life span ≤6 months
2. Considering tumor resection within 6 months
3. Failed CBD cannulation
4. Hilar stricture (Bismuth II, III and IV)
5. CBD dilating by a balloon catheter with diameter≥8mm
6. Inserting the whole FCSEMS into CBD and the distal end of FCSEMS invisible in endoscopic view
7. Maximal CBD diameter ≤6mm
8. Pregnancy or lactation
9. Unable to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
Migration rate of FCSEMS | 6 months
  The proportion of patients who had stent migration after placing FCSEMS, which was defined as radiological or endoscopic evidence of distal or proximal migration within 6 months after placing FCSEMS.

SECONDARY OUTCOMES:
Distal migration rate | 6 months
  The proportion of patients who had distal migration of FCSEMS, which was defined as radiological or endoscopic evidence of fully or partially distal migration of the stent out of CBD during follow up.
  Fully distal migration: The whole stent was out of CBD or disappeared in fluoroscopy.
  Partially distal migration: More than half length of FCSEMS was visible in endoscopic view.
Proximal migration rate | 6 months
  The proportion of patients who had proximal migration of FCSEMS, which was defined as radiological or endoscopic evidence of fully or partially proximal migration of the stent into CBD during follow up.
  Fully proximal migration: The whole stent was in CBD and the distal end was not visible.
  Partially proximal migration: Less than 0.5cm of distal end of FCSEMS was visible in endoscopic view.
Rate of cholangitis after FCSEMS placement | 6 months
  The proportion of patients who had the complication of cholangitis during follow up, due to stent migration, tumor/tissue ingrowth or food impaction.
Complications related to stent removal | 6 months
  Including failed extraction of the stent, bleeding or cholangitis which needed further management after stent removal.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Xiamen Humanity Hospital, Xiamen, Fujian
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi
  - Department of gastroenterology, Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Third Affiliated Hospital of Second Military Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Shi X, Luo H, Ren G, Wang X, Zhao J, Li H, Ning B, Yi H, Zhong L, Zhang R, Ni Z, Liang S, Xia M, Hu B, Pan Y, Fan D. Effects of Clip Anchoring on Preventing Migration of Fully Covered Self-Expandable Metal Stent in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography: A Multicenter, Randomized Controlled Study. Am J Gastroenterol. 2024 Oct 1;119(10):2028-2035. doi: 10.14309/ajg.0000000000002813. Epub 2024 Apr 15. PMID 38619136